CLINICAL TRIAL: NCT03407417
Title: A Patient-centered Intervention Using Technology to Reduce Colorectal Cancer Disparities in Primary Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: IRB201702765 -N; 1R01CA207689-01A1 (NIH); OCR17004 (Other: UF OnCore)
Record Dates: First submitted 2018-01-15; First posted 2018-01-23 (Actual); Results first posted 2025-05-06 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-04

CONDITIONS: Colo-rectal Cancer
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Who Masked: Participant
Masking Description: Study Team will recruit an ethnically diverse sample of eligible patients to complete the intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Human (VH) (Experimental): Patients were randomly assigned to a virtual human (VH) screening condition after completing the eligibility for CRC requirements.
  Interventions: Other: virtual technology
- Text-Base (TB) (Experimental): Patients were randomly assigned to a text-based (TB) screening condition after completing the eligibility for CRC requirements.
  Interventions: Other: virtual technology

INTERVENTIONS:
Other: virtual technology — The app will first ask participants a short series of questions designed to assess their baseline risk for colon cancer. Highly tailored patient reminders will be customized using all 12 constructs.
  Other Names: Virtual human application (ALEX)

SUMMARY:
The purpose of this proposal is to test the efficacy of a patient-centered, tailored message intervention delivered via virtual technology for increasing colorectal cancer (CRC) screening within guidelines among racial/ethnic minority and rural patients. This protocol focuses on the clinical portion of grant NCI 1RCA207689-01A1

DETAILED DESCRIPTION:
Patients will be recruited via a secure, clinical data warehouse to complete a patient-randomized test of the efficacy of the intervention for promoting initial and repeat FIT testing. Patients identified as eligible will be contacted through MyChart to test a web-based, culturally-sensitive virtual human intervention for CRC screening. The web-application will provide information to encourage CRC screening. Therefore, this study is a minimal risk study.

ELIGIBILITY:
Inclusion Criteria:

* able to read English or Spanish at least at eighth-grade level
* have an email account or the ability to receive texts
* willingness to be re-contacted
* consent to MRR related to CRC screening
* not remember completing any CRC screening within recommended guidelines (i.e., <10 years for colonoscopy, <1 year for stool test).
* complete a FIT test:
* a) with a negative result only
* b) complete a FIT test with a positive result AND undergo a completion screening colonoscopy,
* Or c) complete a colonoscopy only.

Exclusion Criteria:

* unable to read English at least at eighth-grade level
* doesn't have an email account or the ability to receive texts
* unwilling to be re-contacted
* Unable to consent to MRR related to CRC screening
* have not had <10 years for colonoscopy, or 1 year for stool test

Ages: 45 Years to 73 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 960 (Actual)
Dates: Start 2018-11-08 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Lok, Principal Investigator — University of Florida
Locations (2):
- United States (2):
  - University of Florida, Gainesville, Florida
  - University of Florida, Jacksonville, Florida

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Virtual Human (VH) Screening: Patients were randomly assigned to a virtual human (VH) screening condition after completing the eligibility for CRC requirements.
  virtual technology - highly tailored VH: The app will first ask participants a short series of questions designed to assess their baseline risk for colon cancer. Highly tailored patient reminders will be customized using all 12 constructs. The VH-tailored content was presented using an animated computer-generated character to deliver tailored, culturally aligned health messages about CRC screening.
- Text-Based (TB) Screening: Patients were randomly assigned to a text-based (TB) screening condition after completing the eligibility for CRC requirements.
  virtual technology - tailored minimally TB: The app will first ask participants a short series of questions designed to assess their baseline risk for colon cancer. Minimally tailored patient reminders will be customized using 4 randomly selected constructs. The TB-tailored content was presented using an image of a computer-generated character to deliver tailored, culturally aligned health messages about CRC screening.
Period: Overall Study
Arm/Group | Virtual Human (VH) Screening | Text-Based (TB) Screening
Started | 482 | 478
Completed | 473 | 470
Not Completed | 9 | 8

BASELINE CHARACTERISTICS:
Population: Although 482 participants were initially enrolled in the Virtual Human (VH) Screening arm and 478 in the Text-Based (TB) Screening arm, only those who completed the baseline assessment were included in the analysis. Specifically, 473 VH participants and 470 TB participants completed the baseline, while 9 and 8 participants, respectively, did not complete it. These 17 individuals were excluded from the analysis due to incomplete baseline data.
Groups:
- Total: Total of all reporting groups
Arm/Group | Virtual Human (VH) Screening | Text-Based (TB) Screening | Total
Number analyzed (Participants) | 473 | 470 | 943
Age, Categorical [Count of Participants; unit: Participants] — Population: Although 482 participants were initially enrolled in the Virtual Human (VH) Screening arm and 478 in the Text-Based (TB) Screening arm, only those who completed the baseline assessment were included in the analysis. Specifically, 473 VH participants and 470 TB participants completed the baseline, while 9 and 8 participants, respectively, did not complete it. These 17 individuals were excluded from the analysis due to incomplete baseline data.
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 381 | 359 | 740
    >=65 years | 92 | 111 | 203
Sex/Gender, Customized [Count of Participants; unit: Participants] — Population: The study did not require participants to self-report their sex. There is no sex data for 40 participants.
  Participants
    Male | 135 | 142 | 277
    Female | 324 | 302 | 626
    Sex not reported | 14 | 26 | 40
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 27 | 26 | 53
  Not Hispanic or Latino | 425 | 411 | 836
  Unknown or Not Reported | 21 | 33 | 54
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 5 | 4 | 9
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 2 | 2 | 4
  Black or African American | 196 | 205 | 401
  White | 240 | 212 | 452
  More than one race | 7 | 13 | 20
  Unknown or Not Reported | 22 | 32 | 54

OUTCOME MEASURES:

1. Primary Outcome: Intention to Screen for Colorectal Cancer (CRC)
Description: Measure: Intention to Screen for Colorectal Cancer Item: I want to get screened for colorectal cancer. Scale: 5-point Likert scale (1 = strongly disagree to 5 = strongly agree). Mean scores near 1 indicate a lower intention to get screened for colorectal cancer. Mean scores near 5 indicate a higher intention to get screened for colorectal cancer.
  Construct: Behavioral intention to screen No subscales
Time Frame: within the first 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Virtual Human (VH) | Text-Base (TB)
Number analyzed (Participants) | 473 | 470
units on a scale | 4.33 (.94) | 4.45 (.86)

2. Secondary Outcome: Communication With a Provider About Colorectal Cancer (CRC)
Description: Measure: Intention to talk to doctor about colorectal cancer screening. Construct: Behavioral intention to communicate Item: I will talk to my healthcare provider about colorectal cancer screening. Scale: 5-point Likert scale (1 = strongly disagree to 5 = strongly agree). Mean scores near 1 indicate a lower intention to talk to a healthcare professional about colorectal cancer screening. Mean scores near 5 indicate a high intention to talk to a healthcare professional about colorectal cancer screening.
  No subscales
Time Frame: Assessed after 24 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Virtual Human (VH) Screening | Text-Based (TB) Screening
Number analyzed (Participants) | 473 | 470
units on a scale | 4.32 (.91) | 4.33 (.90)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for 5 years and 2 months.
Description: During the study, 943 participants were monitored/assessed for other (non-serious) adverse events, but none were observed. We followed a non-systematic method, such as participants' self-reports, to identify whether or not adverse events occurred.
Arm/Group | Virtual Human (VH) Screening | Text-Based (TB) Screening
All-Cause Mortality (participants affected / at risk) | 0/473 | 0/470
Serious Adverse Events (participants affected / at risk) | 0/473 | 0/470
Other Adverse Events (participants affected / at risk) | 0/473 | 0/470

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-11-17): https://cdn.clinicaltrials.gov/large-docs/17/NCT03407417/Prot_SAP_001.pdf
  • Informed Consent Form (2023-10-30): https://cdn.clinicaltrials.gov/large-docs/17/NCT03407417/ICF_000.pdf